CLINICAL TRIAL: NCT02894281
Title: Pupillometry Dynamic Measures in Patients Without Ocular or Neurological Disease
Acronym: PCT
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CLL_2016_2
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Optic Neuritis
Keywords: Pupillary light reflex; Multiple sclerosis
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Measure of pupillary light reflex: patients without optic neuritis
  Interventions: Device: pupillary light reflex
- patients with optic neuritis: clinical database of 22 patients (measurement of pupillary light reflex already performed for the same purpose, in a former study)
  Interventions: Device: pupillary light reflex

INTERVENTIONS:
Device: pupillary light reflex — measure with infra-red cameras

SUMMARY:
Retrobulbar optic neuritis (NORB) is the damage to the optic nerve caused by inflammation. It causes a rapidly progressive and painful visual loss, often among young subjects. Diagnosis confirmation is important to start proper treatment, because a NORB is often the first symptom of multiple sclerosis. This diagnosis, based on a set of arguments, is difficult to define by a non-expert ophthalmologist.

The pupillary light reflex is a way to test the visual afferent pathways. If it is subject to a large inter-individual variability, the dynamics of the pupillary light reflex and its latency are more reproducible. An easy way to study the dynamics of the pupillary light reflex is to study the pupillary cycle time (PCT). In the case of NORB, elongation of the conduction in the visual afferent pathways related to demyelination plate increases the latency of the pupillary light reflex and decreases the frequency of the PCT.

Our hypothesis is that PCT dynamics measures would be a reliable indicator and easy to evaluate some pathologies affecting the integrity of the nerve. The validation of a decrease in the frequency of the PCT in NORB, compared to the frequency observed in subjects ophthalmological or neurological disease, could help developing methods to study the conduction of the visual pathways with portable devices used during the standard ophthalmologic consultation and quickly orientate patients to specialized centers.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* Subject without known ocular or neurological disease
* Ametropia inferior to 3 diopters for spherical correction and inferior to 1.50 diopter for astigmatism correction
* Matched for age and sex with one of the 22 subjects of the patients' unilateral NORB database

Exclusion Criteria:

* history of disease affecting pupillary motility
* anisocoria
* patient under legal protection
* pregnant or breast feeding patient
* patient's refusal to participate in the study
* no medical insurance coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with no optic neuritis are recruited, to be compared with a database of 22 patients already recruited in a former study (measurement of pupillary light reflex already performed in that study, for the same purpose)
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
pupillary cycle time | baseline
  Pupillary cycle time, measured in Hertz

CONTACTS AND LOCATIONS:
Overall Officials: Cedric Lamirel, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France